CLINICAL TRIAL: NCT02344992
Title: Blood Glucose Control With BioChaperone Insulin Lispro Compared to Insulin Lispro (Humalog®) After Ingestion of a Standardized Meal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Adocia (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: BC3-CT011; 2014-005028-92 (EudraCT Number)
Record Dates: First submitted 2015-01-19; First posted 2015-01-26 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2015-06

CONDITIONS: Diabetes Mellitus Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Lispro

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Biochaperone Insulin Lispro (Experimental)
  Interventions: Drug: BioChaperone insulin lispro
- Humalog® (Active Comparator)
  Interventions: Drug: Humalog®

INTERVENTIONS:
Drug: BioChaperone insulin lispro — Single dose of 0.2 U/kg body weight injected subcutaneously
  Arms: Biochaperone Insulin Lispro
Drug: Humalog® — Single dose of 0.2 U/kg body weight injected subcutaneously
  Arms: Humalog®

SUMMARY:
The addition of BioChaperone to already marketed prandial insulin analogue accelerates the onset and shorten the duration of action of insulin lispro due to facilitation of the absorption of the insulin after subcutaneous injection.

This trial is intented to compare the post-prandial blood glucose control of BioChaperone insulin lispro and Humalog® when injected after a standardized meal as well as the pharmacokinetic profile of BioChaperone insulin lispro and Humalog® in subjects with type 1 diabetes mellitus.

This is a double-blinded, randomized, controlled, two-period crossover phase Ib trial to compare the blood glucose control after ingestion of a standardized meal, with BioChaperone Lispro at 0.2U/Kg and Humalog at 0.2U/Kg.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes Mellitus ≥ 12 months
* Treated with multiple daily insulin injections or CSII ≥ 12 months
* BMI 18.5-28.0 kg/m² (both inclusive)
* HbA1C%≤9%

Exclusion Criteria:

* Type 2 Diabetes Mellitus
* Receipt of any trial product within 60 days prior to this trial
* Clinically significant abnormal haematology, biochemistry, lipids or urinalysis screening tests as judged by the investigator considering the underlying disease
* Presence of clinically significant acute gastroinstestinal symptoms as judged by the investigator
* Known slowing of gastric emptying and or gastrointestinal surgery that in the opinion of the investigator might change gastrointestinal motility and food absorption.
* Any systemic treatment with drugs known to interfere with glucose metabolism
* Use of any tobacco or nicotine-contained product within one year prior to screening

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2015-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Area under the blood glucose time curve: AUCbg(0-2h) | 2 hours
  Area under the blood glucose concentration time curve from 0-2 hours after a standardised meal

SECONDARY OUTCOMES:
Pharmacodynamic: Area under the blood glucose concentration time curve from 0-8 hours after a standardized meal: AUCbg(0-8h) | 8 hours
Pharmacodynamic: maximum blood glucose concentration after a standardized meal: BGmax | 8 hours
Pharmacokinetic: Area under the serum insulin lispro concentration time curve from 0-8hours: AUClisp(0-8h) | 8 hours
Pharmacokinetic: Maximum observed serum insulin lispro concentration: Cmax(lisp) | 8 hours
Safety and tolerability: adverse events, local tolerability, vital signs variation, ECG, laboratory safety parameters | Up to 7 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Grit Andersen, MD, Principal Investigator — Profil GmbH
Locations (1):
- Profil GmbH, Neuss, Germany